CLINICAL TRIAL: NCT02072564
Title: Pilot Study on the Influence of the Different Components of the Diet and Different Habits (Tobacco, Alcohol, Physical Exercise, Occupation) Results of IVF-ICSI
Brief Title: Influence of Diet and Lifestyle Factors on the Results of the IVF
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Principal Investigator, Juan Jose Espinos Gomez, MD, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: DYP-HAB-2010-01; Desarrollos y proyectos en RA (Other: DYPRA)
Record Dates: First submitted 2013-09-24; First posted 2014-02-26 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Lifestyle Factors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Couples with indication for IVF: Couples with primary or secondary infertility with indication of IVF
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire with 100 questions divided into different groups: general data, work, physical activity, character, hobbies, disease and diet.

SUMMARY:
The purpose of this study is study the possible relationship between various lifestyle habits of men and women (age, body mass index, diet, exercise, alcohol, tobacco, coffee, etc..) and live birth rate after in vitro fertilization-intracytoplasmatic injection (IVF-ICSI).

DETAILED DESCRIPTION:
It is a prospective study of couples with primary or secondary infertility, with indication for IVF. The main objective is to relate different lifestyle factors (age, BMI, physical activity, tobacco consumption, alchol, drugs, work and diet) with reproductive outcomes obtained in terms of total oocytes, M II, fertilization and implantation rates pregnancy and abortion rates and live birth. It also attempts to correlate the different habits of life in men with seminal parameters. For this, both members of the pair separately should answer a validated questionnaire before beginning the therapeutic process.

ELIGIBILITY:
Inclusion Criteria:

* Couples who want a pregnancy
* Mediterranean or Caucasian Ethnicity.
* Infertility to justify treatment with IVF / ICSI-TEI.
* First cycle of IVF / ICSI.
* Between 18 and 37 years (inclusive)
* Presence of one or both ovaries and uterus can withstand embryo implantation and pregnancy.
* Body mass index (BMI) <40.
* Absence of pregnancy before starting ovarian stimulation.
* Having given their written consent.

Exclusion Criteria:

* Clinically important disease.
* Inclusion in previous cycles of assisted reproduction.
* Unexplained vaginal bleeding.
* Any contraindication to become pregnant.
* Known allergy to preparations of gonadotropins or its excipients.
* Patients undergoing oocyte donation cycles -

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study sample is obtained from the population of infertile couples who meet the criteria for inclusion in a protocol for controlled ovarian stimulation for IVF/ICSI.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Live birth rate | One year

SECONDARY OUTCOMES:
Pregnancy rate | 1 month
Number of mature oocytes | Two weeks
Fertilization rate | Two weeks
Cancelation rate | One month
Total dose | One month
  Total dose of gonadotrophins needed to stimulate the follicular growth
Total Sperm count | Two weeks
  Total number of spermatozoa in the seminal and number of spermatozoa/ml
Abortion rate | 16 weeks
Hyperstimulation rate | One month
  Moderate and severe hyperstimulation

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Espinós-Gómez, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain